CLINICAL TRIAL: NCT03630510
Title: Ventilator Hyperinflation With Increase of Inspiratory Time on Respiratory Mechanics: A Randomized Crossover Trial
Brief Title: Ventilator Hyperinflation With Increase of Inspiratory Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brazilian Institute of Higher Education of Censa (Other)
Responsible Party: Principal Investigator, Luciano Matos Chicayban, Chefe do Laboratório de Análise de Disfunções Pneumofuncionais (LADPF), Brazilian Institute of Higher Education of Censa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VHI + Tins
Record Dates: First submitted 2017-03-02; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Lung Infection; Mechanical Ventilation
Keywords: Physical Therapy Modalities,; Respiration Artificial,; Respiratory Care Units,; Respiratory Mechanics,; Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: The VHI maneuver with inspiratory time adjustment was performed in the pressure controlled ventilation mode (PCV). The inspiratory pressure was increased gradually every 5 cmH2O until reaching a maximum pressure of 35 cmH2O, according to the tolerance of the patient determined by the absence of cough. PEEP remained unchanged throughout the study. The maneuver was performed for 5 min, followed by tracheal aspiration. To perform the control (CTRL), the patients were only positioned and aspirated, without alteration in ventilatory parameters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mechanical ventilator hyperinflation (Experimental): The VHI maneuver with inspiratory time adjustment was performed in the pressure controlled ventilation mode (PCV). The inspiratory pressure was increased gradually every 5 cmH2O until reaching a maximum pressure of 35 cmH2O, according to the tolerance of the patient determined by the absence of cough. PEEP remained unchanged throughout the study. After reaching a maximum pressure of 35 cmH2O (PCV + PEEP level), the inspiratory time was gradually increased until the inspiratory flow reached the baseline. Concomitantly, the respiratory rate was decreased to allow the expiratory flow also to reach the baseline, to avoid self-PEEP. The maneuver was performed for 5 min, followed by tracheal aspiration.
  Interventions: Other: Ventilator hyperinflation
- Control (No Intervention): To perform the control (CTRL), the patients were only positioned and aspirated, without alteration in ventilatory parameters.

INTERVENTIONS:
Other: Ventilator hyperinflation — The ventilator hyperinflation maneuver with inspiratory time adjustment was performed in the pressure controlled ventilation mode (PCV). The inspiratory pressure was increased gradually every 5 cmH2O until reaching a maximum pressure of 35 cmH2O, according to the tolerance of the patient determined by the absence of cough. PEEP remained unchanged throughout the study. After reaching a maximum pressure of 35 cmH2O (PCV + PEEP level), the inspiratory time was gradually increased until the inspiratory flow reached the baseline. Concomitantly, the respiratory rate was decreased to allow the expiratory flow also to reach the baseline, to avoid self-PEEP. The maneuver was performed for 5 min, followed by tracheal aspiration.
  Arms: mechanical ventilator hyperinflation

SUMMARY:
The investigators hypothesis is that the adjustment of the inspiratory time may optimize the distribution of ventilation and increase tidal volume, producing potential therapeutic effects on the displacement of secretions and respiratory mechanics. The objective of this study was To evaluate the effects of hyperinflation with the ventilator associated with increased inspiratory time on respiratory mechanics.

DETAILED DESCRIPTION:
A randomized crossover clinical trial was conducted with 38 mechanically ventilated patients with pulmonary infection. The order of hyperinflation or control (without changes in parameters) was randomized. Hyperinflation was performed for 5 minutes in the controlled pressure ventilation mode, with progressive increases of 5cmH2O until reaching a maximum pressure of 35cmH2O, maintaining PEEP. After reaching 35cmH2O, the inspiratory time and respiratory rate were adjusted so that the inspiratory and expiratory flows reached the baseline, respectively. Static compliance (Cest, sr), total resistance (Rsr) and airway resistance (Rva), slow pressure drop (ΔP2) and peak expiratory flow (PEF) were assessed before (PRÉ), immediately after the maneuver (POSSimed) and after aspiration (POSPasp). Two-way ANOVA was used for repeated measurements with Tukey post-test, considering a significant p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation for more than 48h
* Mucus hypersecretion (defined as the need for suctioning < 2-h intervals)

Exclusion Criteria:

* Severe bronchospasm,
* Positive end expiratory pressure > 10cmH2O,
* PaO2-FiO2 relationship < 150,
* Mean arterial pressure < 60mmHg,
* Pleural effusion or pneumothorax undrained,
* Bronchopleural or tracheoesophageal fistula,
* Decompensated congestive heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Static compliance of respiratory system | Baseline (before), immediately after VHI and five minutes after aspiration
  Compliance was assessed through the occlusion maneuver at the end of inspiration, considering tidal volume, plateau pressure and PEEP. Three measurements were taken at each moment, the mean being used.
Total Resistance of respiratory system | Baseline (before), immediately after VHI and five minutes after aspiration
  The total resistance of the respiratory system was evaluated through the occlusion maneuver at the end of the inspiration, considering the resistive pressure, measured by the difference between the maximum plateau pressure. Three measurements were taken at each moment, the mean being used.
Airway Resistance | Baseline (before), immediately after VHI and five minutes after aspiration
  The airway resistance was assessed by means of the occlusion maneuver at the end of the inspiration, considering the rapid fall of the pressure immediately after the occlusion, measured by the difference between the maximum pressure and P1. Three measurements were taken at each moment, the mean being used.
Peak expiratory flow | Baseline (before), immediately after VHI and five minutes after aspiration
  The peak expiratory flow was evaluated through passive expiration, being considered the greatest value of the flow in the expiratory phase.

CONTACTS AND LOCATIONS:
Overall Officials: LUCIANO M CHICAYBAN, Principal Investigator — Brazilian Institute of Higher Education of Censa
Locations (1):
- Luciano M Chicayban, Campos dos Goytacazes, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chicayban LM. Acute effects of ventilator hyperinflation with increased inspiratory time on respiratory mechanics: randomized crossover clinical trial. Rev Bras Ter Intensiva. 2019 Oct 14;31(3):289-295. doi: 10.5935/0103-507X.20190052. eCollection 2019. PMID 31618346